CLINICAL TRIAL: NCT02524444
Title: A Comparative Study of Mefloquine and Sulphadoxine-pyrimethamine as Prophylaxis Against Malaria in Pregnant Human Immunodeficiency Virus Positive Patients
Brief Title: A Comparative Study of Mefloquine and S-P as Prophylaxis Against Malaria in Pregnant HIV + Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ORIYOMI OMOTOYOSI AKINYOTU (Other)
Collaborators: University of Ibadan (Other)
Responsible Party: Sponsor-Investigator, ORIYOMI OMOTOYOSI AKINYOTU, SENIOR REGISTRAR, University of Ibadan
Organization: University of Ibadan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FDAAA
Record Dates: First submitted 2015-08-05; First posted 2015-08-14 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Malaria in Pregnant HIV + Patients
Keywords: Intermittent preventive therapy; malaria; pregnant; HIV positive; Prevention
MeSH Terms: conditions — Malaria; HIV Seropositivity | interventions — Mefloquine; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mefloquine (Active Comparator): Tabs Mefloquine 250mg 3 doses 4 weeks apart
  Interventions: Drug: Mefloquine
- Sulphadoxine-Pyrimethamine (Active Comparator): 500mg of Sulphadoxine and 25mg of Pyrimethamine 3tablets 4 weeks apart for 3 doses
  Interventions: Drug: Sulphadoxine-Pyrimethamine

INTERVENTIONS:
Drug: Mefloquine — Tabs Mefloquine 250mg
  Other Names: Larimef
  Arms: Mefloquine
Drug: Sulphadoxine-Pyrimethamine — Sulphadoxine 500mg , Pyrimethamine 25mg
  Other Names: Vitadar, Fansidar
  Arms: Sulphadoxine-Pyrimethamine

SUMMARY:
Randomized controlled single blind prospective comparative study.

DETAILED DESCRIPTION:
This study is intended to be a randomized controlled single blind prospective comparative study conducted to compare the efficacy of three, monthly doses of sulphadoxine-pyrimethamine as intermittent preventive therapy with Mefloquine as-intermittent preventive therapy in HIV-infected pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant HIV positive patients
* Gestational age 16 weeks and above
* No history of use of Mefloquine or Sulphadoxine
* Pyrimethamine four weeks prior to recruitment.

Exclusion Criteria:

* Anaemia packed cell volume less than 30%
* Pre -existing medical conditions- Diabetes Mellitus, -Hypertension
* Allergy to Sulphadoxine- Pyrimethamine or Mefloquine
* Non-consenting patients
* Multiple gestation
* Known psychiatric illness
* Known seizure disorder
* History of severe renal or hepatic disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Level of malaria parasitemia in HIV positive women at delivery after administration of Mefloquine or sulphadoxine-pyrimethamine as prophylaxis for malaria in pregnancy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: AYODELE O AROWOJOLU, MBBS IBADAN, Study Director — UNIVERSITY COLLEGE HOSPITAL,IBADAN,OYO STATE, NIGERIA; ORIYOMI O AKINYOTU, MBBS IBADAN, Principal Investigator — UNIVERSITY COLLEGE HOSPITAL,IBADAN,OYO STATE,NIGERIA; ADENIKE F BELLO, MBBS IBADAN, Study Director — UNIVERSITY COLLEGE HOSPITAL,IBADAN,OYO STATE, NIGERIA
Locations (1):
- University College Hospital, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Steketee RW, Wirima JJ, Slutsker L, Khoromana CO, Heymann DL, Breman JG. Malaria treatment and prevention in pregnancy: indications for use and adverse events associated with use of chloroquine or mefloquine. Am J Trop Med Hyg. 1996;55(1 Suppl):50-6. doi: 10.4269/ajtmh.1996.55.50. PMID 8702037
- [Derived] Pons-Duran C, Wassenaar MJ, Yovo KE, Marin-Carballo C, Briand V, Gonzalez R. Intermittent preventive treatment regimens for malaria in HIV-positive pregnant women. Cochrane Database Syst Rev. 2024 Sep 26;9(9):CD006689. doi: 10.1002/14651858.CD006689.pub3. PMID 39324693
- [Derived] Akinyotu O, Bello F, Abdus-Salam R, Arowojolu A. Comparative study of mefloquine and sulphadoxine-pyrimethamine for malaria prevention among pregnant women with HIV in southwest Nigeria. Int J Gynaecol Obstet. 2018 Aug;142(2):194-200. doi: 10.1002/ijgo.12516. Epub 2018 May 25. PMID 29719927